CLINICAL TRIAL: NCT02239835
Title: Tipranavir: An Open-label, Randomized Study Comparing Combination Therapy (Tipranavir and Ritonavir vs. Saquinavir and Ritonavir) Used With Two Nucleoside Reverse Transcriptase Inhibitors in Single Protease Inhibitor-experienced HIV-1 Patients
Brief Title: Tipranavir and Ritonavir vs. Saquinavir and Ritonavir Used With Two Nucleoside Reverse Transcriptase Inhibitors in Single Protease Inhibitor-experienced HIV-1 Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1182.4
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir; Ritonavir; Saquinavir

ARMS (3):
- TPV low dose + RTV low dose (Experimental)
  Interventions: Drug: Tipranavir (TPV) low dose; Drug: Ritonavir low dose
- TPV high dose + RTV low dose (Experimental)
  Interventions: Drug: Tipranavir (TPV) high dose; Drug: Ritonavir low dose
- SQV + RTV high dose (Active Comparator)
  Interventions: Drug: Ritonavir high dose; Drug: Saquinavir

INTERVENTIONS:
Drug: Tipranavir (TPV) low dose
  Arms: TPV low dose + RTV low dose
Drug: Tipranavir (TPV) high dose
  Arms: TPV high dose + RTV low dose
Drug: Ritonavir low dose
  Arms: TPV high dose + RTV low dose; TPV low dose + RTV low dose
Drug: Ritonavir high dose
  Arms: SQV + RTV high dose
Drug: Saquinavir
  Arms: SQV + RTV high dose

SUMMARY:
Objectives of the study were to evaluate the efficacy and safety of two different doses of tipranavir (TPV) in combination with ritonavir (TPV/r) compared with a standard dual PI combination of saquinavir (SQV) and ritonavir (RTV) and to evaluate the dose response of two different doses of TPV in combination with RTV for efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Clinical failure while on the current PI-containing regimen of indinavir, nelfinavir, or amprenavir
* In the investigator's opinion, adherence to the present PI-containing regimen
* Exposure of >=6 months to the current PI therapy
* Stable PI-containing regimen, i.e., receiving the current two reverse transcriptase inhibitors (RTIs) for at least 2 months prior to study entry
* HIV-1 RNA >=1000 copies/mL (assayed using the Amplicor polymerase chain reaction (PCR) method at the initial screening visit)
* No limit in CD4+ cell count at the initial screening
* At least two new nucleoside reverse transcriptase inhibitor (NRTI) options available
* Age >=18 years
* Acceptable screening laboratory test values that indicated adequate baseline organ function at the time of screening. Acceptable laboratory test values consisted of the following: severity <=Grade 1 (ACTG Grading Scale). Stable Grade 2 abnormalities were permitted if the values had been demonstrated and documented for at least >=2 months. All laboratory values >Grade 2 were subject to approval by the P&U Clinical Program Leader or designated personnel and subsequently by the BI designated personnel
* Acceptable medical history, physical examination, ECG, and chest radiograph prior to entry into the treatment phase of the study
* Use of a barrier contraceptive method of birth control for at least 30 days prior to study drug administration, during the study, and 30 days after study completion
* Ability to swallow numerous tablets and capsules without difficulty
* Ability to understand and provide informed consent. Minors had to have approval of a parent or legal guardian

Exclusion Criteria:

* Treatment with more than one PI-containing regimen
* Clinically significant active or acute (onset within the month previous to study entry) medical problems, including the following: opportunistic infections, e.g., active cryptococcosis, Pneumocystis carinii pneumonia, herpes zoster, histoplasmosis, or cytomegalovirus; nonopportunistic diseases, including but not limited to the following: progressive multifocal leukoencephalopathy, lymphoma, or malignancy requiring systemic therapy
* Prior exposure (>7 days) to tipranavir, saquinavir, or ritonavir
* History of clinically significant nervous system or muscle diseases, seizure disorder, or psychiatric disorder that might impair adherence to the protocol
* Taking of any known P450 3A enzyme-inducing drugs within 30 days of study entry and including the following: rifabutin, rifampin, carbamazepine, dexamethasone, phenobarbital, phenytoin, sulfadimidine, sulfinpyrazone, or troleandomycin
* Hypersensitivity to tipranavir, saquinavir, or ritonavir
* Use of interferons, interleukins, HIV vaccines, or any active immunizations within 30 days of study entry
* Taking of any investigational medication with the exception of adefovir dipivoxil (Preveon™) within 30 days of study entry
* Pregnancy or lactation (serum β-human chorionic gonadotrophin test had to have been negative within 14 days of study entry)
* Evidence of substance abuse, which in the investigator's opinion could affect adherence to the protocol
* In the investigator's judgment, inability to comply with the protocol requirements for reasons other than those specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 1999-12; Primary Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in plasma HIV-1 RNA concentrations | Week 16, 24 and 48
Occurrence of HIV-1 RNA levels below the limit of quantitation (BLQ) | up to 96 weeks
  using the Roche Amplicor HIV Monitor™ Method [limit of detection (LD) 400 copies/mL] and the Roche Amplicor UltraSensitive Method™ (LD 50 copies/mL)
Number of patients with treatment-emergent and drug-related adverse events (AEs) | up to 96 weeks
Number of patients with serious adverse events (SAEs) | up to 96 weeks
Number of patients with grade 3 and 4 laboratory abnormalities | up to 96 weeks

SECONDARY OUTCOMES:
Change from baseline in cluster of differentiation (CD) 4+ cell count | Week 16, 24 and 48
Time to virologic failure | after week 16
  defined as plasma HIV-1 RNA values >400 copies/mL at two consecutive time points 2 to 4 weeks apart
Occurrence of new or recurring AIDS-defining illnesses | up to 96 weeks
Occurrence of HIV-1 related illness | up to 96 weeks
Occurrence of death | up to 96 weeks
Time to new or recurring AIDS-defining illnesses | up to 96 weeks
Time to HIV-1 related illness | up to 96 weeks
Time to death | up to 96 weeks
Change from baseline in blood glucose | up to 96 weeks
Change from baseline in cholesterol | up to 96 weeks
Change from baseline in high density lipoprotein (HDL) | up to 96 weeks
Change from baseline in triglycerides | up to 96 weeks
Time to virologic response | up to 96 weeks
Trough plasma tipranavir concentrations | up to week 24
Sequence-based HIV-1 analysis (genotyping) and drug susceptibility assays (phenotyping) | Baseline and week 24